CLINICAL TRIAL: NCT05139927
Title: Using the Multiphase Optimization Strategy (MOST) to Optimize an Intervention to Increase COVID-19 Testing for Black and Latino/Hispanic Frontline Essential Workers
Brief Title: Using MOST to Optimize an Intervention to Increase COVID-19 Testing for Frontline Essential Workers
Acronym: NCAP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY2022-6023
Record Dates: First submitted 2021-11-29; First posted 2021-12-01 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; COVID-19 Testing
Keywords: multiphase optimization strategy (MOST); COVID-19 testing; Black and Latino; frontline essential workers
MeSH Terms: conditions — COVID-19 | interventions — Motivational Interviewing; Counseling

STUDY DESIGN:
Intervention Model Description: Full factorial experiment testing 4 behavioral intervention components. There are 16 conditions needed to test the effects of the 4 components. Each condition comprises a combination of components. In the sections that follow, we describe the 16 conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - ON Component C: Peer education - ON Component D: Navigation
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 2 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - ON Component C: Peer education - ON Component D: Self-test kit
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 3 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - ON Component C: Peer education - ON Component D: Navigation
  Interventions: Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 4 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - ON Component C: Peer education - ON Component D: Self-test kit
  Interventions: Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 5 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - OFF Component C: Peer education - ON Component D: Navigation
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 6 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - OFF Component C: Peer education - ON Component D: Self-test kit
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 7 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - OFF Component C: Peer education - ON Component D: Navigation
  Interventions: Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 8 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - OFF Component C: Peer education - ON Component D: Self-test kit
  Interventions: Behavioral: Peer education; Behavioral: Access to COVID testing
- Condition 9 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - ON Component C: Peer education - OFF Component D: Navigation
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Access to COVID testing
- Condition 10 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - ON Component C: Peer education - OFF Component D: Self test kit
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Access to COVID testing
- Condition 11 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - ON Component C: Peer education - OFF Component D: Navigation
  Interventions: Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Access to COVID testing
- Condition 12 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - ON Component C: Peer education - OFF Component D: Self test kit
  Interventions: Behavioral: Text messages (TMs) and quiz questions (QQs); Behavioral: Access to COVID testing
- Condition 13 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - OFF Component C: Peer education - OFF Component D: Navigation
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Access to COVID testing
- Condition 14 (Experimental): Component A: motivational interviewing counseling - ON Component B: Text message intervention - OFF Component C: Peer education - OFF Component D: Self test kit
  Interventions: Behavioral: Motivational interviewing (MI) counseling; Behavioral: Access to COVID testing
- Condition 15 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - OFF Component C: Peer education - OFF Component D: Navigation
  Interventions: Behavioral: Access to COVID testing
- Condition 16 (Experimental): Component A: motivational interviewing counseling - OFF Component B: Text message intervention - OFF Component C: Peer education - OFF Component D: Self test kit
  Interventions: Behavioral: Access to COVID testing

INTERVENTIONS:
Behavioral: Motivational interviewing (MI) counseling — Those assigned to receive Component A will engage in a MI single session lasting approximately 30-45 minutes. The overall goal of the session is to increase participants' motivation and readiness to test for COVID-19 in various circumstances.
  Arms: Condition 1; Condition 10; Condition 13; Condition 14; Condition 2; Condition 5; Condition 6; Condition 9
Behavioral: Text messages (TMs) and quiz questions (QQs) — This intervention lasts 6 weeks. This component is grounded in principles of behavioral economics. Its main goal is to add interest and excitement to the goal of COVID-19 testing, serve as a reminder that COVID-19 testing is recommended in a number of scenarios, and "nudge" participants toward testing and creating a habit of serial screening and COVID-19 testing as needed. Participants first receive a brief orientation to the component (15 min.), and the participant will put the study phone number into his/her phone and a test TM and QQ will be sent. TMs and QQs are programmed into the Telerivet program and sent automatically. Twice a week participants will receive a TM with information about COVID and COVID-19 testing followed by a true/false question about that TM two days later, for which they earn 10 points for a correct answer, and 5 points for an incorrect answer. Participants earn modest prizes based on their points.
  Arms: Condition 1; Condition 10; Condition 11; Condition 12; Condition 2; Condition 3; Condition 4; Condition 9
Behavioral: Peer education — This component has two aspects: Participants are trained to educate their peers on core messages about the importance of COVID-19 testing that address social norms about COVID-19 testing and highlight COVID-19 testing as an altruistic act (15-20 min. training). Then, participants are given the opportunity to educate three peers who are Black and Latino/Hispanic frontline essential workers on the core messages. These peers contact the study directly and receive a brief assessment and referrals to testing, but are not enrolled in the study.
  Arms: Condition 1; Condition 2; Condition 3; Condition 4; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Access to COVID testing — Component D is an adaptive intervention component that avoids unnecessary costs; it is only provided if needed. Level 1: Over a 2-3 week period, navigation includes a brief needs assessment and guidance to assist participants in prioritizing, accessing, and completing COVID-19 testing sequences in a timely fashion and resolving barriers such as transportation or the possible need to take off work if diagnosed with COVID-19. Level 2: 1 month after enrollment, participants will be contacted by phone. If they have not been tested, we will provide them with a BinaxNOW test kit which can be picked up or mailed to them.

SUMMARY:
COVID-19 testing is essential to controlling the COVID-19 pandemic to break transmission chains and reduce community transmission. However, Black and Latino/Hispanic populations in lower status frontline essential occupations such as food preparation, retail, building maintenance, personal services, and in-home health care have serious barriers to COVID-19 testing and, therefore, insufficient testing rates. The proposed study will use the multiphase optimization strategy framework to address the problem of low COVID-19 testing rates for this population: We will test the effects of four distinct candidate intervention components and then create an efficient multicomponent made up of the most effective combination of the components that can be rapidly scaled up in community settings to boost COVID-19 testing rates.

DETAILED DESCRIPTION:
The proposed study responds to RFA-OD-21-008 which calls for community-engaged interventions to support COVID-19 testing in underserved and vulnerable populations. Among those at highest risk for exposure to COVID-19 is the large population of frontline essential workers (FEW) in lower status occupations (e.g., retail, in-home health care), among whom Black and Latino/Hispanic (BLH) persons are over-represented. The CDC recommends testing for all those experiencing symptoms of COVID-19. For those not vaccinated, testing is recommended after exposure to individuals with a COVID-19 diagnosis, and regular COVID-19 screening testing is recommended even when asymptomatic for those with frequent close contact with others in indoor settings such as FEW. However, BLH-FEW experience serious impediments to COVID-19 testing at individual/attitudinal- (e.g., lack of knowledge of guidelines, distrust), social- (e.g., social norms), and structural-levels of influence (e.g., poor access to testing). Indeed, testing rates are lower among BLH than White populations and only 25-50% of BLH-FEW are currently vaccinated. The proposed community-engaged study is led by a collaborative team at New York University and the Northern Manhattan Improvement Corporation (NMIC). Its main goal is to optimize a behavioral intervention to boost COVID-19 testing rates for BLH-FEW. Consistent with RFA-OD-21-008, the proposed study uses the multiphase optimization strategy (MOST) framework to test four candidate intervention components grounded in our past research. The candidate components are informed by critical race theory and guided by the theory of triadic influence, are brief or do not require substantial staff time, and will be tested in a highly efficient factorial experimental design. They are A) motivational interview counseling, B) a text message component grounded in behavioral economics, C) peer education, and D) access to testing (via navigation to a test appointment vs. a self-test kit). All participants receive the standard of care, namely, health education on COVID-19 testing, and referrals. The specific aims of the study are to: identify which of four candidate components contribute meaningfully to improvement in the primary outcome, COVID-19 testing with medical confirmation; the most effective combination of components will comprise the "optimized" intervention (Aim 1), identify mediators (e.g., distrust, access) and moderators (e.g., sociodemographic characteristics) of the effects of each component (Aim 2), and use a mixed-methods approach to explore relationships among barriers to, facilitators of, and uptake of COVID-19 testing and COVID-19 vaccination (Aim 3). Participants will be N=448 BLH-FEW who have not been tested for COVID-19 in the past three months and have not been vaccinated for COVID-19 in the past 12 months, randomly assigned to an intervention condition, and assessed at 6- and 12-weeks post-baseline; N=50 participants will engage in qualitative in-depth interviews. We will also uncover, describe, and plan for implementation issues so the optimized intervention can be rapidly scaled up by NMIC and other community-based organizations.

ELIGIBILITY:
INCLUSION CRITERIA: 1) age 18-70 years; 2) can engage in study activities in English or Spanish; 3) Black or African American (including Caribbean, African, or multi-ethnic Black) and/or Latino or Hispanic race/ethnicity; 4) resides in NYC; 5) in the past month, was employed as a frontline worker in a lower status essential occupation in one or more of the domains listed above; 6) has a phone that can be used for study participation and can receive TMs; 7) has not received any doses of a COVID-19 vaccination in the past 12 months; 8) has not been tested for COVID-19 in the past three months; 9) if previously diagnosed with COVID-19, has not been symptomatic in the past two weeks or 90 days has passed since treatment with monoclonal antibodies or convalescent plasma98; 10) has not been educated/interviewed as a peer for Component C; 11) willing to engage in a core session and be randomly assigned to receive 1-4 components.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marya Gwadz, PhD, Principal Investigator — New York University
Locations (1):
- New York University Silver School of Social Work, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gwadz M, Cleland CM, Lizardo M, Hawkins RL, Bangser G, Parameswaran L, Stanhope V, Robinson JA, Karim S, Hollaway T, Ramirez PG, Filippone PL, Ritchie AS, Banfield A, Silverman E. Using the multiphase optimization strategy (MOST) framework to optimize an intervention to increase COVID-19 testing for Black and Latino/Hispanic frontline essential workers: A study protocol. BMC Public Health. 2022 Jun 21;22(1):1235. doi: 10.1186/s12889-022-13576-0. PMID 35729622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The optimization randomized controlled trial described here was conducted in New York City between July 2022 and February 2024. The trial was a collaboration between New York University and the Northern Manhattan Improvement Corporation. Study activities were conducted at a research field site in lower Manhattan. Persons could participate there in-person or engage in the study virtually. Recruitment took place in the community,
Groups:
- Condition 1: Component A: MIC - ON Component B: TM - ON Component C: PE- ON Component D: Navigation
Period: Overall Study
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
Started | 24 | 28 | 28 | 27 | 26 | 28 | 28 | 28 | 27 | 28 | 28 | 28 | 27 | 28 | 28 | 27
Completed | 24 | 28 | 28 | 27 | 26 | 28 | 28 | 28 | 27 | 28 | 28 | 28 | 27 | 28 | 28 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Information is the same
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16 | Total
Number analyzed (Participants) | 24 | 28 | 28 | 27 | 26 | 28 | 28 | 28 | 27 | 28 | 28 | 28 | 27 | 28 | 28 | 27 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.46 (10.56) | 36.07 (8.73) | 33.54 (10.12) | 39.44 (12.07) | 35.19 (11.18) | 35.29 (9.56) | 33.82 (9) | 31.82 (8.46) | 35.37 (7.75) | 36.04 (11.44) | 35.64 (9.19) | 35.54 (10.07) | 32.59 (8.66) | 33.89 (9.32) | 34.75 (9.16) | 32.41 (9.11) | 34.93 (9.65)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self report: What terms best express how you describe your gender identity? (SELECT ONE)
  Responses: woman, man, non-binary, transgender man, transgender woman, none, other
  Note that we had missing data on sex assigned at birth so we relied on gender for this study. In most cases, sex and gender are the same.
  Participants
    Man/male gender | 8 | 12 | 20 | 15 | 15 | 16 | 12 | 16 | 12 | 14 | 14 | 19 | 13 | 16 | 13 | 14 | 229
    Female/woman or gender minority | 16 | 16 | 8 | 12 | 11 | 12 | 16 | 12 | 15 | 14 | 14 | 9 | 14 | 12 | 15 | 13 | 209
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black or bi- or multi-racial | 11 | 11 | 15 | 13 | 15 | 12 | 15 | 18 | 10 | 16 | 12 | 12 | 13 | 11 | 17 | 13 | 214
  Other race | 13 | 17 | 13 | 14 | 11 | 16 | 13 | 10 | 17 | 12 | 16 | 16 | 14 | 17 | 11 | 14 | 224
  Latino/Hispanic (yes) | 13 | 17 | 13 | 14 | 11 | 16 | 13 | 10 | 17 | 12 | 16 | 16 | 14 | 17 | 11 | 14 | 224

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Testing at Follow-up Assessment
Description: COVID-19 testing at the 6- and/or 12-week follow-up assessment (at least one instance)
Time Frame: by the 12-week FU
Population: participants
Measure: Mean (Standard Deviation); unit: proportion of those tested at least once
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
Number analyzed (Participants) | 24 | 28 | 28 | 27 | 26 | 28 | 28 | 28 | 27 | 28 | 28 | 28 | 27 | 28 | 28 | 27
proportion of those tested at least once | 0.85 (0.37) | 0.61 (0.5) | 0.63 (0.49) | 0.81 (0.4) | 0.68 (0.48) | 0.59 (0.5) | 0.54 (0.51) | 0.64 (0.49) | 0.64 (0.49) | 0.79 (0.41) | 0.69 (0.47) | 0.68 (0.48) | 0.54 (0.51) | 0.81 (0.4) | 0.56 (0.51) | 0.71 (0.46)

ADVERSE EVENTS:
Time Frame: 12-week follow-up
Description: Several mechanisms were put in place to monitor potential adverse events that participants may experience throughout the study, whether related to project participation or not. Events were classified as Reportable, Adverse, or Not Harmful/Expectable and reported to the IRB and Program Official as required. No adverse events were observed during the study period.
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28 | 0/28 | 0/27 | 0/26 | 0/28 | 0/28 | 0/28 | 0/27 | 0/28 | 0/28 | 0/28 | 0/27 | 0/28 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28 | 0/28 | 0/27 | 0/26 | 0/28 | 0/28 | 0/28 | 0/27 | 0/28 | 0/28 | 0/28 | 0/27 | 0/28 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28 | 0/28 | 0/27 | 0/26 | 0/28 | 0/28 | 0/28 | 0/27 | 0/28 | 0/28 | 0/28 | 0/27 | 0/28 | 0/28 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT05139927/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT05139927/ICF_000.pdf